CLINICAL TRIAL: NCT04932148
Title: The INCremental Dialysis to Improve Health Outcomes in People Starting Haemodialysis (INCH-HD) Study: a Randomised Controlled Trial
Brief Title: INCremental Dialysis to Improve Health Outcomes in People Starting Haemodialysis (INCH-HD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: Medical Research Future Fund (Other); Queensland Health (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AKTN 20.04
Record Dates: First submitted 2021-06-08; First posted 2021-06-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-03

CONDITIONS: Kidney Failure
Keywords: Incremental HD; Incident HD
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incremental HD (Experimental): Participants randomised to incremental HD will commence HD twice weekly and continue until an indication for an increase to three sessions/week (trigger point) is reached.
  Interventions: Other: Incremental HD
- Conventional HD (Other): Participants randomised to conventional HD will commence HD thrice weekly from the first HD session.
  Interventions: Other: Conventional HD

INTERVENTIONS:
Other: Incremental HD — Starting haemodialysis at twice weekly frequency
  Arms: Incremental HD
Other: Conventional HD — Starting haemodialysis at thrice weekly frequency
  Arms: Conventional HD

SUMMARY:
The INCH-HD trial will test if incremental HD preserves the quality of life of patients and families and is a safe, practical, cost effective treatment option.

DETAILED DESCRIPTION:
Kidney failure is a growing public health problem and fatal unless treated with dialysis or transplantation. Haemodialysis is the most common treatment for kidney failure in Australia and globally. Patients find haemodialysis extremely burdensome due to symptoms like fatigue, pain, cramps and poor quality of life that generally equates to <60% of full health. Furthermore, haemodialysis is associated with an extremely high mortality (<50% survive 5 years), particularly in the first 3-6 months of starting haemodialysis, which is likely linked to the rapid loss of patients' own kidney function when starting haemodialysis abruptly at three sessions/week. Observational studies suggest that starting haemodialysis incrementally at two sessions/ week is associated with lower mortality and better preservation of patients' remaining kidney function while offering many patient-important advantages, including dialysis free time and ability to work. However, robust evidence to recommend this incremental approach is lacking.

The INCH-HD study is an investigator-initiated, international, multicentre, prospective, adaptive, randomised, open-label, parallel group, non-inferiority trial. The primary objective of the study is to demonstrate whether incremental HD is non-inferior to conventional HD for the patient-important outcome of quality of life measured using Kidney-specific component of the Kidney Disease Quality of Life - Short Form measurement (KDQOL-SF) at 6 months from dialysis commencement.

The study will recruit a total of 372 participants across HD centres in Australia, and Canada. The outcomes of this trial will will provide urgently needed high quality evidence on whether starting haemodialysis incrementally at two sessions/week compared to the conventional three sessions/week can safely reduce the physical, financial and quality-of life burden on patients, lower early mortality rates and slow loss of kidney function while increasing haemodialysis capacity and reducing costs.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥ 18 years of age) and
2. Commencing HD as their initial dialysis therapy and
3. Able to give informed consent

Exclusion Criteria:

1. Urine output <0.5Litres/day
2. Unlikely to be on HD for ≥1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Heath related quality of life | 6 months
  This will be measured using Kidney-specific component (KSC) of the Kidney Disease Quality of Life Short Form (KDQOL-SF) V1.3 questionnaire. The KSC is the mean of the 11 domains of the kidney-disease specific items of KDQOL-SF. Scores are transformed onto a 0-100 range, where a higher score reflects a better quality of life.

SECONDARY OUTCOMES:
Residual kidney function (RKF) | Baseline, 3, 6, 12 and 18 months
  Calculated as (creatinine clearance + kidney urea clearance) divided by 2 then corrected for body surface area using the DuBois method (0.20247 x (height in centimetres x 0.725) x (weight in kilograms x 0.425).
  Expressed as millilitres per minute (ml/min). Expected range 1 ml/min to 20 ml/min, where lower values indicate worse kidney function.
Healthcare resource utilisation | Baseline to 18 months
  Healthcare resource use over 18 months using linked data and patient monthly calendars
Healthcare costs | Baseline to 18 months
  Healthcare costs over 18 months using linked data and patient monthly calendars
Heath related quality of life using Kidney Disease Quality of Life Short Form (KSQOL-SF) questionnaire | Baseline, 3, 6, 9, 12, 15 and 18 months
  Heath-related quality of life will be measured using Kidney-specific component (KSC) of the Kidney Disease Quality of Life Short Form (KDQOL-SF) V1.3 questionnaire. The KSC is the mean of the 11 domains of the kidney-disease specific items of KDQOL-SF. Scores are transformed onto a 0-100 range, where a higher score reflects a better quality of life.
Heath related quality of life using EuroQol 5-dimension 5-level (EQ-5D-5L) questionnaire | Baseline, monthly to 18 months
  Heath-related quality of life will be measured using EuroQol 5 Domain 5 Level (EQ-5D-5L) questionnaire. EQ-5D has descriptive and visual analogue scale (VAS). Descriptive system consists of five dimensions mobility, self-care, usual activities, pain/discomfort and anxiety/depression. VAS records patient's self-rated health on vertical visual analogue scale with endpoints best to worst health with 0 being worst and 100 being best health.
Incidence of all-cause mortality | Baseline to 18 months
  Incidence of all-cause mortality up to 18 months
Time to major cardiovascular event (MACE) | Baseline to 18 months
  Time to first major cardiovascular event (MACE) up to 18 months
Number of non-elective hospital admissions | Baseline to 18 months
  Number of non-elective hospital admissions up to 18 months
Total hospital days | Baseline to 18 months
  Total hospital days up to 18 months
Time to death | Baseline to 18 months
  Time to death up to 18 months
Number of hospital admissions | Baseline to 18 months
  Number of hospital admissions up to 18 months
Adverse events and side-effects | Baseline to 18 months
  This will include episodes of hyperkalaemia, extra dialysis sessions for fluid overload, number of vascular access complications
Symptom scores | Baseline, 3, 6, 9, 12, 15 and 18 months
  This will be measured using change in the physical and mental component summaries of the Kidney Disease Quality of Life Short Form (KDQOL-SF) V1.3 questionnaire. This is scored using the mean of the physical and mental components of the KDQOL-SF. Scores are transformed onto a 0-100 range, where a higher score reflects a better quality of life.
Fatigue | Baseline, 3, 6, 9, 12, 15 and 18 months
  This will be measured using the Standardised Outcomes in Nephrology-Haemodialysis (SONG-HD) Fatigue questionnaire. The SONG-HD Fatigue measure consists of three items that assess the effect of fatigue on life participation, tiredness, and level of energy. The overall score for fatigue is obtained by summing the responses across the three questions, resulting in a scale ranging from zero (no fatigue) to nine (maximum fatigue).
Nutritional Status | Baseline, 6, 12 and 18 months
  This will be measured using the Subjective Global Assessment (SGA) of nutrition which is scored as proportion of well nourished (A) versus malnourished (B or C). A (well nourished), B (mildly-moderately malnourished), C (Severely malnourished)
Vascular access | Baseline to 18 months
  This will be measured as mumber of functional vascular access interventions required per patient per year to enable and /or maintain vascular access for HD per patient-year

OTHER OUTCOMES:
Patient lifestyle and wellbeing | Baseline, 3, 6, 9, 12, 15 and 18 months
  This will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) SF 4a (Ability to Participate in Social Roles and Activities and Satisfaction with Social Roles and Activities)
Time to event | Baseline to 18 months
  Time to trigger condition being met in Incremental HD patients (date the trigger condition/s were met) and subsequent time to transition to 3x/week HD

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kerr, Prof, Principal Investigator — University of Queensland, Monash University; David Johnson, Prof, Principal Investigator — University of Queensland, Queensland Health; Andrea Viecelli, Dr, Principal Investigator — University of Queensland, Queensland Health; Charmaine Lok, Prof, Principal Investigator — University Health Network, Toronto
Locations (16):
- Australia (15):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Northern Beaches Hospital, Frenchs Forest, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Bundaberg Hospital, Bundaberg, Queensland
  - Cairns Hospital, Cairns, Queensland
  - Redland Hospital, Cleveland, Queensland
  - Logan Hospital, Logan City, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Health, Melbourne, Victoria
  - Eastern Health, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- University Health Network- University of Toronto, Toronto, Ontario, Canada